CLINICAL TRIAL: NCT05403710
Title: Targeting Nociceptors in Hidradenitis Suppurativa
Brief Title: Botulinum Toxin Therapy in Hidradenitis Suppurativa
Acronym: HS
Status: Recruiting | Type: Observational
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Hidradenitis Suppurativa Foundation (Unknown); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Sarah Whitley, Assistant Professor of Dermatology, University of Massachusetts, Worcester
Other Study IDs: STUDY00000805; 7K08AR080844-02 (NIH)
Record Dates: First submitted 2022-05-16; First posted 2022-06-03 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Hidradenitis Suppurativa; Hyperhidrosis
MeSH Terms: conditions — Hidradenitis Suppurativa; Hyperhidrosis | interventions — Botulinum Toxins; Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1. Formalin fixed paraffin embedded (FFPE) skin specimens will be stored at room temperature in dermatopathology clinical specimen bank in a deidentified manner for upto 5 years.
  2. OCT-embedded or snap frozen skin tissue will be stored at -80 degrees celsius in research lab space in a deidentified manner for upto 5 years.
  3. RNA derived from skin tissue will be stored at -80 degrees celsius in research lab space in a deidentified manner for upto 5 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- single group assignment: men or women between the ages of 18-75 who have an established diagnosis of Hidradenitis Suppurativa
  Interventions: Drug: Botulinum toxin

INTERVENTIONS:
Drug: Botulinum toxin — Administration of botulinum toxin (50 units/100cm2 injected intradermally) into lesional skin
  Other Names: Botox

SUMMARY:
This study will build on data from mice and humans implicating TRPV1 nociceptors in the pathogenesis of the type-17 chronic inflammatory skin disease Hidradenitis Suppurativa (HS). In this study, the investigators will test the hypothesis that inhibiting neuropeptide activity with botulinum toxin reduces pathogenic inflammation.

DETAILED DESCRIPTION:
Botulinum toxin prevents vesicle fusion at nerve terminals thereby inhibiting neuropeptide release. The investigators will collect punch biopsies of lesional skin from HS patients before, and 1-2 months after botulinum toxin treatment (50U per axilla in 10 injections of 0.1mL) then perform flow cytometric, transcriptomic, and microscopic analysis of skin to determine if nonselective inhibition of neuropeptide release diminishes IL-17 driven skin inflammation.

ELIGIBILITY:
Inclusion:

* Adults between ages 18 and 75 years with established diagnosis of hidradenitis suppurativa (HS)
* HS skin lesions of duration at least 1 year, HS skin lesions in at least two different body areas

Exclusion:

* Age < 18 years or > 75 years
* pregnant or breastfeeding
* neuromuscular disorder (ex. ALS, myasthenia gravis, Lambert-Eaton syndrome, myopathy)
* medical co-morbidity that is a relative contraindication to skin biopsy procedure (ex. end stage congestive heart failure or coagulopathy)
* active bacterial, fungal, or viral infection in the treatment area
* known hypersensitivity to botulinum toxin A preparations or any of their components (human albumin, saline, lactose, sodium succinate)
* prisoners
* adults unable to consent for themselves.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of men or women between the ages of 18-75 who have an established diagnosis of Hidradenitis Suppurativa who will undergo botulinum toxin treatment as part of routine care.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-06-07 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Quantification and phenotyping of skin resident dendritic cell, macrophage, and T cell populations in patients before and after intralesional Botox treatment. | 1-2 months after first treatment
  immune cell phenotyping

CONTACTS AND LOCATIONS:
Overall Officials: Sarah K Whitley, MD PhD, Principal Investigator — Assistant Professor of Dermatology
Locations (1):
- University of Massachusetts Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Research team will share data and samples from this study with other investigators who are interested in skin diseases, but in that case no patient identifying information will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: for up to 7 years following data collection
Access Criteria: Proposals should be directed to sarah.whitley@umassmed.edu.To gain access to data, requesters will have to sign a data access agreement.

REFERENCES:
- [Background] Campanati A, Martina E, Giuliodori K, Bobyr I, Consales V, Offidani A. Two cases of Hidradenitis suppurativa and botulinum toxin type a therapy: A novel approach for a pathology that is still difficult to manage. Dermatol Ther. 2019 May;32(3):e12841. doi: 10.1111/dth.12841. Epub 2019 Feb 10. PMID 30693648
- [Background] Shih T, Lee K, Seivright JR, De DR, Shi VY, Hsiao JL. Hyperhidrosis treatments in hidradenitis suppurativa: A systematic review. Dermatol Ther. 2022 Jan;35(1):e15210. doi: 10.1111/dth.15210. Epub 2021 Nov 30. PMID 34796606
- [Background] Grimstad O, Kvammen BO, Swartling C. Botulinum Toxin Type B for Hidradenitis Suppurativa: A Randomised, Double-Blind, Placebo-Controlled Pilot Study. Am J Clin Dermatol. 2020 Oct;21(5):741-748. doi: 10.1007/s40257-020-00537-9. PMID 32761500
- [Background] Campanati A, Martina E, Giuliodori K, Consales V, Bobyr I, Offidani A. Botulinum Toxin Off-Label Use in Dermatology: A Review. Skin Appendage Disord. 2017 Mar;3(1):39-56. doi: 10.1159/000452341. Epub 2017 Feb 1. PMID 28612001
- [Background] Kimball AB, Sobell JM, Zouboulis CC, Gu Y, Williams DA, Sundaram M, Teixeira HD, Jemec GB. HiSCR (Hidradenitis Suppurativa Clinical Response): a novel clinical endpoint to evaluate therapeutic outcomes in patients with hidradenitis suppurativa from the placebo-controlled portion of a phase 2 adalimumab study. J Eur Acad Dermatol Venereol. 2016 Jun;30(6):989-94. doi: 10.1111/jdv.13216. Epub 2015 Jul 22. PMID 26201313
- [Background] Kim YS, Hong ES, Kim HS. Botulinum Toxin in the Field of Dermatology: Novel Indications. Toxins (Basel). 2017 Dec 16;9(12):403. doi: 10.3390/toxins9120403. PMID 29258169